CLINICAL TRIAL: NCT02746471
Title: Medtronic Reveal LINQ Insertable Cardiac Monitor Registry
Brief Title: Reveal LINQ Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Reveal LINQ Registry
Record Dates: First submitted 2016-02-29; First posted 2016-04-21 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-03

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Reveal LINQ

SUMMARY:
The Reveal LINQ Registry will generate reliable long-term "real world" data of product performance, economic valuation, site-of-service procedural information.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, observational, multi-center, global study. The study will characterize clinical actions initiated by Reveal LINQ arrhythmia detection and estimate procedure-related acute infection rate. Approximately 1,500 subjects will be implanted with a Reveal LINQ ICM and undergo continuous remote monitoring and be followed prospectively from insertion through 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements.
* Subject is intended to receive or be treated with the have a Reveal LINQ ICM inserted in the next 30 days.
* Patient enrolled before or on the same date of insertion of the Reveal LINQ ICM
* Subject consent prior to ICM insertion

Exclusion Criteria:

* Subject who is, or is expected to be inaccessible for follow-up
* Subject with exclusion criteria required by local law
* Subject is currently enrolled in or plans to enroll a concurrent study that may confound the results of this study. Co-enrollment in any concurrent drug and/or device clinical study (including registries) requires approval of the study manager or designee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to receive a market-released Reveal LINQ device are eligible to enroll in the Registry. All enrolled patients that have an attempted procedure will be included in the analysis. Consented patients who failed to receive a Reveal LINQ device may be exited from the registry when all reportable events are resolved.
Sampling Method: Non-Probability Sample
Enrollment: 1604 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, M.D., Principal Investigator — The Valley Hospital
Locations (48):
- United States (19):
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Jacksonville Heart (Baptist Medical), Jacksonville, Florida
  - Bay Heart Group, Tampa, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - NYU Langone Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute (Dallas-TX), Dallas, Texas
  - Baylor Research Institute (Fort Worth TX), Fort Worth, Texas
  - Baylor Research Institute (Plano TX), Plano, Texas
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Ziekenhuis Oost Limburg - Campus St.-Jan, Leuven, Belgium
- Evaggelismos Hospital, Athens, Greece
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - Ospedale classificato ed equiparato Sacro Cuore, Negrar
  - Presidio Ospedaliero Santa Maria del Carmine, Rovereto
- Japan (14):
  - National Kyushu Medical Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Hirosaki University Hospital, Hirosaki
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kyorin University Hospital, Mitaka
  - Iwate Medical University Hospital, Morioka
  - Okayama University Hospital, Okayama
  - Ogaki Municipal Hospital, Ōgaki
  - Showa University Hospital, Shinagawa-Ku
  - National Cerebral and Cardiovascular Center, Suita
  - The Jikei University School of Medicine Hospital, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Fujita Health University Hospital, Toyoake
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht Universitair Medisch Centrum (MUMC), Maastricht
- Portugal (6):
  - Centro Hospitalar Lisboa Ocidental - Hospital de Santa Cruz, Carnaxide
  - Hospital Senhora da Oliveira, Guimaraes, Guimarães
  - Centro Hospitarlar Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Hospital do Espirito Santo, Ponta Delgada
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto
  - Hospital Distrital de Santarem, Santarém
- Saudi Arabia (2):
  - King Fahd Armed Forces Hospital, Jeddah
  - Prince Sultan Cardiac Center, Riyadh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beinart SC, Natale A, Verma A, Amin A, Kasner S, Diener HC, Del Greco M, Wilkoff BL, Pouliot E, Franco N, Mittal S. Real-world comparison of in-hospital Reveal LINQ insertable cardiac monitor insertion inside and outside of the cardiac catheterization or electrophysiology laboratory. Am Heart J. 2019 Jan;207:76-82. doi: 10.1016/j.ahj.2018.10.002. Epub 2018 Oct 14. PMID 30487072

RESULTS

PARTICIPANT FLOW:
Groups:
- Registry: 1604 subjects were enrolled in the study from 55 centers in US, EMEA and Saudi Arabia.
  Follow-up data collection ended on 04 Jun 2021.
Period: Overall Study
Arm/Group | Registry
Started | 1604
Completed | 442
Not Completed | 1162
Not completed — Death | 43
Not completed — Exited before 36 months | 1119

BASELINE CHARACTERISTICS:
Population: Subjects who had a LINQ device implanted.
Groups:
- LINQ Subjects: Subjects who were confirmed to have been implanted with a LINQ device
Arm/Group | LINQ Subjects
Number analyzed (Participants) | 1604
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 770
  >=65 years | 806
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 682
  Male | 922
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 233
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 47
  White | 877
  More than one race | 10
  Unknown or Not Reported | 435
Region of Enrollment [Number; unit: participants]
  Greece | 32
  Saudi Arabia | 42
  Netherlands | 41
  Belgium | 35
  United States | 920
  Japan | 215
  Italy | 166
  Israel | 8
  Portugal | 101
  Germany | 27
  United Kingdom | 6
  Spain | 11
NYHA [Count of Participants; unit: Participants] — New York Heart Association (NYHA) classification for the stages of Heart Failure. Values range from I-IV. Higher values indicate more severe limitations in patient activity due to symptoms
  Participants
    Class I | 27
    Class II | 27
    Class III | 9
    Not Available | 195
    Patient does not have Heart Failure | 1346
Reason for Implant [Count of Participants; unit: Participants]
  AF Management | 177
  Cryptogenic Stroke | 291
  Palpitations | 177
  Post-AF Ablation Monitoring | 78
  Pre-AF Ablation Monitoring | 27
  Seizures | 2
  Suspected AF | 178
  Syncope | 540
  Transient Ischemic Attack (TIA) | 9
  Ventricular Tachycardia | 49
  Other | 76

OUTCOME MEASURES:

1. Primary Outcome: Number and Type of Clinical Actions Initiated by Reveal LINQ Arrhythmia Detection Feature
Description: Clinical actions taken over the course of study follow-up
Time Frame: Implant to 36 months post-implant
Population: Subjects who had an opportunity to have an action taken after ICM insertion
Measure: Number; unit: Number of times action taken
Arm/Group | Registry
Number analyzed (Participants) | 1604
Number of times action taken
  AF Ablation | 201
  Electrical Cardioversion | 75
  Other Ablation | 32
  PCI | 9
  PFO Closure | 4
  Therapeutic Device Implanted | 176
  Aortic valve replacement | 1
  Placement of a Watchman device | 1
  Stopped OAC medication at least once during study (was on at baseline) | 141
  Started OAC medication at least once during study (was off at baseline) | 176

2. Primary Outcome: Number of Participants With Procedure-related Acute Infection Rate
Description: Acute infection rate in the subjects who were followed for at least 30 days or had an infection prior to 30 days. Infections are as assessed by the Investigator and defined as deep incision site or superficial infection.
  Deep incision site are classified as pain, redness, or drainage at incision site requiring the device to be removed or IV antibiotics administered.
  Superficial infections are defined as redness beyond procedure expectation and oral antibiotics administered.
  For both deep incision and superficial infections, a physician directed intervention must occur for the event to be defined as an infection.
Time Frame: Implant to 30 days post-implant
Population: Same as arm/group description
Measure: Count of Participants; unit: Participants
Groups:
- Safety Cohort: Subject was enrolled in the study prior to their Reveal LINQ insertion and the subject either completed at least one visit at a time point ≥ 30 days post insertion procedure or the subject had an infection event reported on or prior to 30 days.
Arm/Group | Safety Cohort
Number analyzed (Participants) | 1261
Participants | 8

ADVERSE EVENTS:
Time Frame: Up to 36 months of study enrollment
Description: Systematic Assessment: At follow-up visits subjects were asked about occurrence of adverse events.
Arm/Group | Registry
All-Cause Mortality (participants affected / at risk) | 43/1604
Serious Adverse Events (participants affected / at risk) | 64/1604
Other Adverse Events (participants affected / at risk) | 0/1604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Registry (N=1604)
Cerebrovascular accident (Nervous system disorders) | 15 (16)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Device expulsion (Product Issues) | 1 (1)
Device extrusion (Product Issues) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 3 (3)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Pocket erosion (Injury, poisoning and procedural complications) | 4 (5)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 8 (8)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PI's may not publish single-site data until the main multi-site publication has occurred.

DOCUMENTS (2):
  • Study Protocol (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02746471/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02746471/SAP_001.pdf